CLINICAL TRIAL: NCT03287076
Title: A Multicentre, Randomised Controlled Trial of Exenatide Versus Standard Care in Acute Ischemic Stroke (TEXAIS)
Brief Title: Trial of EXenatide in Acute Ischaemic Stroke
Acronym: TEXAIS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Neuroscience Trials Australia (Other)
Collaborators: National Health and Medical Research Council, Australia (Other); Monash University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NTA1127; 2018-004325-88 (EudraCT Number)
Record Dates: First submitted 2017-07-13; First posted 2017-09-19 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Acute Ischemic Stroke
Keywords: stroke; glucose; exenatide
MeSH Terms: conditions — Ischemic Stroke; Stroke | interventions — Exenatide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Active (Experimental): Patients will receive exenatide injections
  Interventions: Drug: Exenatide Injection
- Standard Care (No Intervention): Standard care for stroke as per hospital protocol

INTERVENTIONS:
Drug: Exenatide Injection — 5μg subcutaneously twice daily for five days, commencing within 9 hours of symptom onset
  Other Names: Byetta
  Arms: Active

SUMMARY:
A multicentre, randomised controlled Trial of Exenatide versus standard care in Acute Ischemic Stroke

DETAILED DESCRIPTION:
Overview: Elevated blood glucose levels are common in many acute diseases, resulting in worse clinical outcomes. Hyperglycaemia in acute ischaemic stroke (post-stroke hyperglycaemia [PSH]) occurs in up to 50% patients, reduces the efficacy of stroke thrombolysis with increased risk of haemorrhage, increases infarct size, and results in worse clinical outcomes and death. Insulin-based therapies have not proved beneficial in treating PSH: they are difficult to implement and maintain, cause frequent hypoglycaemia, may cause increased infarct size, and do not reduce mortality or improve clinical outcomes. An alternative, simple to use, treatment for PSH may therefore have a significant impact not only for acute stroke care, but in other acute diseases.

Pilot data: Exenatide is a commonly used diabetes drug (a synthetic glucagon- like peptide-1 receptor agonist) that increases insulin secretion. Importantly, this action is glucose dependent - as blood glucose levels decrease, its stimulatory effect on insulin secretion subsides, with a very low risk of hypoglycaemia. A small randomised pilot study of 17 consecutive, unselected patients (ie. regardless of their admission glucose level) with acute ischaemic stroke compared subcutaneous exenatide 5μg for 5 days with routine standard of care. Overall, blood glucose levels remained consistently lower (and less variable) in the exenatide group, and most noticeably in those stroke patients with known diabetes. Exenatide was safe and well tolerated by all patients, with no symptomatic hypoglycaemia.

Trial design: TEXAIS is a 3 year Phase 2, multi centre, prospective, randomised, open label, blinded end-point (PROBE) trial comparing Exenatide to Standard of Care. The sample size is 528 patients (264 in each arm).

Intervention: Treatment arm will receive Exenatide (Byetta) 5μg subcutaneously twice daily for five days, commencing within 9 hours of symptom onset. Stroke onset time for wake-up strokes is taken as mid-point between going to bed, and waking up. Antiemetic therapy (metoclopramide or ondansetron) will be commenced with the first dose of Exenatide. In patients receiving tPA, Exenatide will be given alongside, or as soon as possible, following tPA administration (within 60 minutes). Diabetic patients already on oral agents and/or insulin may continue these (as per standard practice) in addition to Exenatide. Continuous glucose monitors (CGMs) will track the intra-day dynamic variability of glucose in acute stroke.

Translation: TEXAIS is a simple, practical, study that can enrol all patients with ischaemic stroke, regardless of admission blood glucose level, regardless of stroke severity, with no target glucose level, and with low risk of hypoglycaemia.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 18 years or older
* Acute Ischaemic Stroke - CT brain exclusion of haemorrhagic stroke
* Blood glucose level on admission ≥ 4mmol/L
* First trial treatment possible within 9 hours of stroke onset
* Pre-morbid /mRS score of 0-2

Exclusion Criteria:

* Haemorrhagic stroke
* Poor clinical prognosis /palliation (considered unlikely to survive beyond 14 days post stroke).
* Any known allergy or hypersensitivity to Exenatide
* Females who are pregnant (known or suspected) or currently breastfeeding
* Any past history of pancreatitis or evidence of active pancreatitis
* History of active severe gastrointestinal disease (including but not limited to gastroparesis and dumping syndrome)
* Current chronic kidney disease stage 4 or 5 (creatinine clearance <30ml/min)
* Current participation in another interventional clinical trial
* Inability to provide consent (participant or person responsible as local laws apply)
* Current use of Exenatide (Byetta®), or other GLP-1 agonist diabetes medication
* Patients considered unlikely to be able to be followed up at 3 months (including but not limited to geographical location of patient at 3 months)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2017-11-23 (Actual); Primary Completion 2021-10-04 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
improved neurological outcome | 7 days
  Treatment with short acting Exenatide (Byetta) in patients with acute ischaemic stroke is hypothesised to improve neurological outcome as measured by ≥8 point improvement in the National Institutes of Health Stroke Scale (NIHSS) stroke disability score (or NIHSS 0-1) at 7 days

SECONDARY OUTCOMES:
post stroke hyperglycaemia | 90 days
  reduce the occurrence of post stroke hyperglycaemia (>7mmol/l).
Modified Rankin Scale | 90 days
  improve Modified Rankin Scale (mRS) at 90 days
NIHSS | 90 days
  improve NIHSS at 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Bladin, Principal Investigator — The Florey Institute of Neuroscience & Mental Health Melbourne Brain Centre
Locations (15):
- Australia (13):
  - St Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Sunshine Coast University Hospital, Birtinya, Queensland
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Launceston General Hospital, Launceston, Tasmania
  - Box Hill Hospital, Box Hill, Victoria
  - St Vincent's Hospital Melbourne, Fitzroy, Victoria
  - Austin Hospital, Heidelberg, Victoria
  - Alfred Hospital, Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - St John of God Midland Public & Private Hospital, Midland, Western Australia
  - Fiona Stanley Hospital, Murdoch, Western Australia
- Helsinki University Hospital, Helsinki, Finland
- CDHB Christchurch Hospital, Christchurch, New Zealand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bladin CF, Wah Cheung N, Dewey HM, Churilov L, Middleton S, Thijs V, Ekinci E, Levi CR, Lindley R, Donnan GA, Parsons MW, Meretoja A, Tiainen M, Choi PMC, Cordato D, Brown H, Campbell BCV, Davis SM, Cloud G, Grimley R, Lee-Archer M, Ghia D, Sanders L, Markus R, Muller C, Salvaris P, Wu T, Fink J; TEXAIS Investigators. Management of Poststroke Hyperglycemia: Results of the TEXAIS Randomized Clinical Trial. Stroke. 2023 Dec;54(12):2962-2971. doi: 10.1161/STROKEAHA.123.044568. Epub 2023 Nov 27. PMID 38011235